CLINICAL TRIAL: NCT02834910
Title: Prevalence, Characterization and Risk Factors of Acquiring Qnr Genes in Extended Spectrum Beta-lactamase Producing Enterobacteriaceae Isolated in East Inter-region.
Brief Title: Qnr Genes in Enterobacteriaceae
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 173IR08
Record Dates: First submitted 2016-07-13; First posted 2016-07-15 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Enterobacteriaceae Infection
MeSH Terms: conditions — Enterobacteriaceae Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Case group: patients with Extended-Spectrum Beta-lactamase producing Enterobacteriaceae carrying a qnr gene isolate
  Interventions: Other: collection of bacterial sample
- control-group: patients with Enterobacteriaceae isolate without qnr gene
  Interventions: Other: collection of bacterial sample

INTERVENTIONS:
Other: collection of bacterial sample

SUMMARY:
Enterobacteriaceae are bacteria of the gastrointestinal tract which are also the most frequently involved in bacterial infections, especially urinary tract infections. Because of their presence in the gut, these bacteria are the most exposed to antibiotic treatment administered to patients.

Therefore, many antibiotic resistance mechanisms are observed in some of them. Quinolone antibiotics are often used because of their distribution in the body, of the great number of bacterial species that are sensitive to these antibiotics and the possibility to give oral treatments.

For a long time no transferable resistance gene to quinolones from one bacterium to another had been observed. This phenomenon has been demonstrated in 1998 in a bacterium of the Klebsiella pneumoniae species carrying a qnrA gene which encodes a protein that protects the target of the antibiotic in the bacteria. Since several genes have been observed. These genes reduce the sensitivity of the bacteria without ever reach detectable resistance levels on the tests commonly used in the laboratory. However, these genes are often found among enterobacteria in combination with other mechanisms of resistance to other classes of antibiotics including beta-lactam antibiotics that are widely used antibiotics.

Moreover, it is considered that quinolone administration to bacteria carrying these qnr genes could promote the emergence of mutants resistant to quinolones to a more high-level. That furthers multiresistance emergence when the bacteria is already resistant to beta-lactam antibiotics.

The aim of this study performed between April 2008 and March 2009 was to collect strains resistant to beta-lactams because of the production of enzymes, called extended-spectrum beta-lactamase to determine quinolone resistance gene frequency in these bacteria.

Meanwhile, control patients were selected to seek the emergence of these genes risk factors.

The clinical study failed to identify specific risk factors, however, the biological study enhanced the knowledge on this issue with the setting-up of a method for rapid detection of these plasmidic mediated quinolones resistance genes and the description a new plasmid containing a qnr gene, qnrD, whose study is still ongoing.

DETAILED DESCRIPTION:
The multidrug resistance in Enterobacteriaceae is a recurring concern for the treatment of patients. Given their epidemic character, the bacteria that produce extended spectrum beta-lactamase (ESBLs) are subject to extensive and costly preventive measures. Gene location of the first described ESBL were plasmids which could transfer from one species to another often associated with resistance to aminoglycoside. Quinolone resistance was not transferable. In 1998, was discovered a Klebsiella pneumoniae carrying a qnr A plasmid gene encoding a protein protecting girases and topoisomerase IV against quinolones. Yet the levels of ciprofloxacin MIC achieved by strains harboring this gene without any other quinolones resistance mechanism associated, remain low. However, the ciprofloxacin MICs for Escherichia coli lacking any other quinolone resistance mechanism can go from 0.003 mg / L to 0.25 mg / L, depending on the type of qnr. Currently, three types of qnr genes have been described, encoding proteins having several variants (qnrA (n = 6), qnrB (n = 10) and qnrS (n = 2). The qnrA and qnrB genes are carried by plasmids of 54-180 kb. Gene environment on plasmid DNA is that of class 1 integron or Type sul1 called. However the sequenced plasmids carrying qnrS do not have integron-like structures. These genes are more common in the Enterobacteriaceae strains producing ESBL strains than in the others. The low prevalences observed up to date, are increasing in some studies. We have observed qnr in 9 of 138 (6.5%) strains isolated in Champagne-Ardenne in 2004, including 4 of 10 strains of Enterobacter cloacae. Furthermore it has been shown in vitro that the presence of qnrA gene facilitated mutant selection for high-level quinolone resistance. Therefore, given the increasing trend in the prevalence of this gene reported by some authors, it is necessary to establish a monitoring and identify factors favoring the emergence of these strains. The purpose of the study is to observe the evolution of the prevalence of qnr genes within ESBL-producing strains, to detect the emergence of an epidemic clonal strain, and look for the emergence of risk factors of these genes. Given the low prevalence of these genes that research involves a multicenter study which will be organized on 9 East region's inter hospitals from 1 April 2008 to 31 March 2009. It is therefore a descriptive study that clinicobiological aims to: - To collect a sufficient number of producer strains of these genes, - To characterize their different variants (CHU Reims), - To identify the clones possibly associated with these genes (Besançon University Hospital), - To study their genetic environment (CHU Dijon), - Seek clinical factors and antibiotic treatments favoring their presence. All ESBL-producing Enterobacteriaceae isolates, identified in the 5 CHU inter region and CH 4, Colmar, Vesoul, Troyes and Charleville for one year will be centralized at the Bacteriology Laboratory of the University Hospital of Reims. The non duplicate isolates will be included (one isolate per patient resistance phenotype, by species and by month). 600 ESBL-producing strains are expected in this period and among them 50 strains carrying the gene qnr. The clinical study is a retrospective record. For each patient with a isolate carrying qnr, 2 control patients from the same hospital with an age difference of less than 10 years with the "case" will be drawn in the list of patients who had a ESBL producing Enterobacteriaceae. And 150 patient records will be included in the study. Parallel sequencing of qnr genes will allow their precise identification and highlight variants. The quinolones MICs will be determined to detect any increase in the level of resistance. The rest of the study include ESBL identification by sequencing. The study of the genetic environment of qnr will be performed for one isolate by gene type and by species for detecting genetic factors promoting their dissemination (plasmid, integron), variabilities compared to the literature data and get additional epidemiological markers. Genotyping of the isolates will highlight a possible epidemic clone. For Escherichia coli phylogenetic group will be determined at the University Hospital of Besancon. The distribution of E. coli strains. coli carrying the qnr among different phylogenetic groups will be compared to that of a number of isolates of Escherichia coli drawn among the ESBL strains having no qnr (2 controls for 1 case). The major clinical parameters recorded from the files will be, among others, the reason for hospitalization, the main underlying disease, antibiotic treatment before and after the isolation of ESBL bacteria. It will determine if the strains carrying the gene qnr are statistically more resistant to certain molecules that stem not having.

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized

Exclusion Criteria:

* <18 yo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For one year, plasmidic mediated quinolone resistance (PMQR) were detected all the Extended- Spectrum beta-lactamase producing Enterobacteriaceae isolated in the 5 teaching hospitals and 4 general hospitals of the french East inter region during the first nine months of 2009. A case-control study was performed. The cases were the 29 patients in whom a qnr gene was detected in an enterobacteriaceae. The controls were 104 patients hospitalized in the hospital with a age difference < 10 years with a case and having an Enterobacteriaceae without a qnr gene. At least, 2 control patients were selected. for each case
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2009-01; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
number of ESBL-producing strains | 22 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, France, Reims, France